CLINICAL TRIAL: NCT03669887
Title: A Randomized Clinical Trial Using a Postnatal Lifestyle Modification Program to Improve Diet, Adiposity and Metabolic Outcome in Mothers With Gestational Diabetes and Their Offspring
Brief Title: Lifestyle Modification to Improve Diet in Women With GDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Prince of Wales Hospital, Shatin, Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Ronald C.W. Ma, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017.268-T
Record Dates: First submitted 2018-09-12; First posted 2018-09-13 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-02

CONDITIONS: Gestational Diabetes; Diabetes; Childhood Obesity; Diabetes Mellitus
Keywords: Gestational diabetes; Diabetes; Lifestyle; Diet Modification; Childhood Obesity; Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus; Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: In the pilot study that preceded a similar postpartum intervention trial, in which the intervention included telephone counselling (Ferrara et al. 2011). The proportion of women from the control arm who reached the postpartum weight goal was 30%, with the absolute difference in percentage of women meeting the postpartum weight goals being 16% between the intervention and control arms. Assuming a larger between group difference of 20% based on our more intensive individual-level intervention, and a similar 30% of women in the control arm reaching postpartum weight goal, a sample size of 220 (110 in each arm) would give 90% power to detect the between group difference of 20%. Allowing for up to 30% drop-out at 12 months, we planned to recruit 157 subjects in each arm (total sample size n=314).
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle Modification Program (Experimental): Women randomised into the intervention group received the 1-year lifestyle modification program.
  Interventions: Behavioral: Lifestyle Modification Program
- Control (No Intervention): Women randomised into the control arm received standard postnatal care.

INTERVENTIONS:
Behavioral: Lifestyle Modification Program — The intervention will consist of 5 individual face-to-face sessions at 2-weekly intervals with a dietitian with experience in lifestyle modification program, followed by monthly phone contact and smartphone text messages. All study participants in the intervention arm will also be arranged to meet with an exercise instructor at least once during the LMP on the same day as one of the dietitian appointment. Ongoing support from the exercise instructor will also be available by phone calls or emails.
  Arms: Lifestyle Modification Program

SUMMARY:
The study aims to adapt a lifestyle modification program to engage GDM women early in the postnatal period to evaluate its effectiveness in reducing adiposity and metabolic parameters in the mother. Women will be randomized to receive a structured intervention or standard care.

DETAILED DESCRIPTION:
A complex intervention based on a proven lifestyle modification program (LMP) will be delivered to participants randomized to the intervention arm, starting in the early postnatal period. The intervention will consist of individualized face-to-face counseling on diet and weight management, meeting with exercise instructor, followed by telephone contact.

Control will receive standard postnatal education materials and usual care provided by government health service.

ELIGIBILITY:
Inclusion Criteria:

1. Women who developed gestational diabetes in their most recent pregnancy
2. GDM is diagnosed according to the WHO 2013 criteria of FBG ≥ 5.1mmol/l, or 1 hour glucose ≥10.0mmol/l, or 2 hour glucose ≥ 8.5mmol/l during 75g OGTT performed at 24-28 weeks of pregnancy
3. Singleton pregnancy
4. Reside normally in Hong Kong
5. Able to communicate in Chinese
6. Willing to give consent and follow study procedures

Exclusion Criteria:

1. Subjects with pre-existing diabetes (T1D or T2D)
2. Subjects with life-threatening conditions including malignancy that is not in remission
3. Subjects with known psychiatric conditions including depression
4. Substance abuse or use of illicit substances
5. Subjects with significant renal impairment (eGFR<60ml/min at baseline) or non-diabetic renal disease (e.g. biopsy-proven glomerulonephritis or obstructive uropathy)
6. Subjects on chronic corticosteroids treatment
7. Subjects with known myocardial infarction within the preceding 3 months
8. Major physical disability
9. Participation in other intervention trials
10. Surgical or medical interventions to treat obesity
11. Pregnancy at any point during the intervention period

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women had GDM history
Enrollment: 103 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Proportion achieving body weight goal | Baseline, 12 months
  3% body weight change at 12 months if pre-pregnant BMI ≥ 23kg/m2, or for those with pre-pregnant BMI <23 kg/m2, either back to pre-pregnant weight or maintaining within BMI <23 kg/m2

SECONDARY OUTCOMES:
Change in diabetes risk | Baseline, 12 months
  Measured by a validated risk score calculator (RUBY- Risk Understanding By Yourself)
Changes in fasting glucose | Baseline, 12 months
  Measured by OGTT (changes in mmol/l)
Changes in physical activity | Baseline, 12 months
  Measured by International Physical Activity Questionnaires (IPAQ) Total 7 questions on physical activity frequency according to intensity of the physical activity. Higher score indicates more physical activity.
Changes in quality of life indices | Baseline, 12 months
  Measured by Patient Health Questionnaire (PHQ-9) total score 27. Higher score indicates greater severity of depression. (Depression Severity: 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe.)
% of achieving dietary intervention goal | Baseline, 8weeks, 12 months
  Measured by a 3-day food intake record

CONTACTS AND LOCATIONS:
Overall Officials: Ronald C Ma, MBBChir,FRCP, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hosptial, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
We will decide on whether to make data available based on study results and the requests received.

REFERENCES:
- [Background] Tam WH, Ma RC, Yang X, Ko GT, Lao TT, Chan MH, Lam CW, Cockram CS, Chan JC. Cardiometabolic risk in Chinese women with prior gestational diabetes: a 15-year follow-up study. Gynecol Obstet Invest. 2012;73(2):168-76. doi: 10.1159/000329339. Epub 2011 Dec 16. PMID 22179684
- [Background] Tam WH, Ma RC, Yang X, Ko GT, Tong PC, Cockram CS, Sahota DS, Rogers MS, Chan JC. Glucose intolerance and cardiometabolic risk in children exposed to maternal gestational diabetes mellitus in utero. Pediatrics. 2008 Dec;122(6):1229-34. doi: 10.1542/peds.2008-0158. PMID 19047239
- [Background] Tam WH, Ma RCW, Ozaki R, Li AM, Chan MHM, Yuen LY, Lao TTH, Yang X, Ho CS, Tutino GE, Chan JCN. In Utero Exposure to Maternal Hyperglycemia Increases Childhood Cardiometabolic Risk in Offspring. Diabetes Care. 2017 May;40(5):679-686. doi: 10.2337/dc16-2397. Epub 2017 Mar 9. PMID 28279981
- [Background] Woo J, Sea MM, Tong P, Ko GT, Lee Z, Chan J, Chow FC. Effectiveness of a lifestyle modification programme in weight maintenance in obese subjects after cessation of treatment with Orlistat. J Eval Clin Pract. 2007 Dec;13(6):853-9. doi: 10.1111/j.1365-2753.2006.00758.x. PMID 18070255
- [Background] Wong VW, Chan RS, Wong GL, Cheung BH, Chu WC, Yeung DK, Chim AM, Lai JW, Li LS, Sea MM, Chan FK, Sung JJ, Woo J, Chan HL. Community-based lifestyle modification programme for non-alcoholic fatty liver disease: a randomized controlled trial. J Hepatol. 2013 Sep;59(3):536-42. doi: 10.1016/j.jhep.2013.04.013. Epub 2013 Apr 23. PMID 23623998
- [Background] Ferrara A, Hedderson MM, Albright CL, Ehrlich SF, Quesenberry CP Jr, Peng T, Feng J, Ching J, Crites Y. A pregnancy and postpartum lifestyle intervention in women with gestational diabetes mellitus reduces diabetes risk factors: a feasibility randomized control trial. Diabetes Care. 2011 Jul;34(7):1519-25. doi: 10.2337/dc10-2221. Epub 2011 May 3. PMID 21540430